CLINICAL TRIAL: NCT06760065
Title: A Multicenter, Randomized Controlled Study Comparing Keverprazan Hydrochloride-Amoxicillin Dual Therapy and Susceptibility-Guided Quadruple Therapy in Helicobacter Pylori Rescue Treatment
Brief Title: Comparison of Keverprazan Hydrochloride-Amoxicillin Dual Therapy and Susceptibility-Guided Quadruple Therapy for Helicobacter Pylori Rescue Treatment
Acronym: KHDT-SGT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Guangzhou First People's Hospital (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Longgang District People's Hospital of Shenzhen (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other); Bao'an District People's Hospital of Shenzhen (Unknown); Foshan Fuxing Chancheng Central Hospital (Unknown)
Responsible Party: Principal Investigator, Xiang Peng, Attending Physician, Department of Gastroenterology, The Sixth Affiliated Hospital of Sun Yat-Sen University, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHDT-SGT; 1010-Program (Other: The Sixth Affiliated Hospital of Sun Yat-Sen University Clinical Research)
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Helicobacter Pylori Infection Helicobacter Pylori Eradication Patient Education
Keywords: Helicobacter pylori; Keverprazan Hydrochloride; Susceptibility-guided therapy
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: This study uses a parallel design, where participants are randomly assigned to one of two groups: (1) Keverprazan Hydrochloride combined with Amoxicillin as a dual therapy, or (2) a susceptibility-guided quadruple therapy. Each group will receive the assigned treatment independently, and outcomes will be compared to assess the efficacy and safety of both regimens. Randomization ensures balanced allocation, and the parallel model allows for direct comparison of the two interventions under controlled conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Keverprazan Hydrochloride + Amoxicillin (Experimental): Participants in this arm will receive Keverprazan Hydrochloride 20 mg twice daily and Amoxicillin 0.75 g four times daily for 14 days. This dual therapy aims to evaluate the efficacy of Keverprazan Hydrochloride, a potassium-competitive acid blocker, in combination with Amoxicillin for Helicobacter pylori eradication.
  Interventions: Drug: Keverprazan Hydrochloride tablets + high dose amoxicillin
- Susceptibility-Guided Quadruple Therapy (Active Comparator): Participants will receive susceptibility-guided quadruple therapy based on H. pylori resistance testing:
  Clarithromycin-sensitive strains: Esomeprazole 20 mg, Bismuth Potassium Citrate 220 mg, Amoxicillin 1 g, and Clarithromycin 500 mg, twice daily for 14 days.
  Metronidazole-sensitive strains: Esomeprazole 20 mg, Bismuth Potassium Citrate 220 mg, Amoxicillin 1 g, and Metronidazole 400 mg, twice daily for 14 days.
  Levofloxacin-sensitive strains: Esomeprazole 20 mg, Bismuth Potassium Citrate 220 mg, Amoxicillin 1 g (twice daily), and Levofloxacin 500 mg (once daily) for 14 days.
  Multi-drug resistant strains: Esomeprazole 20 mg, Bismuth Potassium Citrate 220 mg, Amoxicillin 1 g, and either Furazolidone 0.1 g (twice daily) or Tetracycline 500 mg (four times daily) for 14 days.
  For Amoxicillin-resistant strains, antibiotics will be adjusted based on susceptibility testing.
  Interventions: Drug: Susceptibility-Guided Quadruple Therapy

INTERVENTIONS:
Drug: Keverprazan Hydrochloride tablets + high dose amoxicillin — Keverprazan Hydrochloride, a potassium-competitive acid blocker (P-CAB), is administered at a dose of 20 mg twice daily in combination with Amoxicillin 0.75 g four times daily for 14 days. This dual therapy is designed to provide rapid and sustained gastric acid suppression and evaluate its efficacy in eradicating Helicobacter pylori.
  Arms: Keverprazan Hydrochloride + Amoxicillin
Drug: Susceptibility-Guided Quadruple Therapy — Participants in this arm will receive quadruple therapy tailored to individual H. pylori resistance profiles, including a proton pump inhibitor (Esomeprazole 20 mg), Bismuth Potassium Citrate 220 mg, and two antibiotics selected based on susceptibility testing (e.g., Amoxicillin, Clarithromycin, Metronidazole, Levofloxacin, or Furazolidone). The regimen is administered for 14 days to optimize eradication outcomes.
  Arms: Susceptibility-Guided Quadruple Therapy

SUMMARY:
This study aims to evaluate the efficacy and safety of Keverprazan Hydrochloride combined with Amoxicillin in dual therapy compared to susceptibility-guided quadruple therapy in the treatment of Helicobacter pylori (H. pylori) infections requiring rescue therapy. H. pylori is a common infectious disease associated with peptic ulcers, gastric cancer, and mucosa-associated lymphoid tissue lymphoma. However, the increasing resistance of H. pylori to antibiotics has reduced the eradication rates of standard therapies.

Potassium-competitive acid blockers (P-CABs), such as Keverprazan Hydrochloride, provide faster and more sustained gastric acid suppression compared to traditional proton pump inhibitors (PPIs), making them a promising option for H. pylori treatment. This multicenter, randomized controlled trial will provide critical evidence comparing the effectiveness of Keverprazan-based dual therapy to susceptibility-guided quadruple therapy, aiming to establish optimized rescue therapy guidelines for H. pylori eradication.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is a globally prevalent chronic infectious disease with an infection rate exceeding 50%. As a Gram-negative bacterium, H. pylori survives in the acidic gastric environment and is a major cause of peptic ulcers, gastric mucosa-associated lymphoid tissue lymphoma, and gastric cancer. Eradication of H. pylori can prevent the recurrence of peptic ulcers and reduce the risk of developing gastric cancer. However, increasing antibiotic resistance has significantly decreased the eradication rate of standard triple therapy to below 80%, posing a substantial challenge to effective H. pylori management.

This study focuses on evaluating a novel potassium-competitive acid blocker (P-CAB), Keverprazan Hydrochloride, in combination with Amoxicillin as dual therapy for H. pylori rescue treatment. P-CABs, including Keverprazan, offer rapid and sustained gastric acid suppression independent of CYP2C19 polymorphism, overcoming limitations of traditional proton pump inhibitors (PPIs). Recent studies have demonstrated the efficacy of P-CABs in first-line H. pylori treatment with high eradication rates and fewer side effects. However, evidence for their use in rescue therapy is currently lacking.

This multicenter, randomized controlled trial aims to compare the efficacy and safety of Keverprazan Hydrochloride-Amoxicillin dual therapy with susceptibility-guided quadruple therapy in patients requiring rescue treatment. The trial will involve patients with confirmed H. pylori infection who failed previous treatment regimens. The study's primary outcome is the eradication rate, and secondary outcomes include the incidence of adverse events and patient compliance.

This research is expected to provide critical evidence for the clinical application of Keverprazan Hydrochloride in H. pylori rescue therapy, potentially establishing it as an effective and patient-friendly treatment option.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged ≥18 years and ≤75 years at the time of signing the informed consent.
2. Participants who have undergone at least one prior standard H. pylori eradication treatment but failed.
3. Current H. pylori infection confirmed by 13C-UBT, or H. pylori culture.
4. Participants who, in the investigator's opinion, are able to understand and comply with the study requirements.
5. Written informed consent and any required privacy authorization documents signed and dated before the initiation of any study procedures.
6. For women of childbearing potential with regular or potential sexual activity with non-sterilized male partners, agreement to use two effective methods of contraception from the time of informed consent until the end of the study.

Exclusion Criteria:

1. Presence of gastric or duodenal ulcer with current or recent bleeding as evidenced by endoscopy.
2. Confirmed gastric cancer by endoscopic biopsy.
3. Receipt of any investigational drug (including marketed drugs used in post-marketing studies) within 30 days prior to the screening period. Participants who failed screening and did not receive the investigational drug may be included.
4. Participants who are investigators, relatives of investigators, or otherwise have conflicts of interest or may be under pressure to participate.
5. History of cutaneous or systemic lupus erythematosus.
6. Clinical manifestations of upper or lower gastrointestinal bleeding within 4 weeks prior to randomization.
7. Diagnosis of Zollinger-Ellison syndrome or other gastric acid hypersecretory disorders.
8. Known allergy or hypersensitivity to Keverprazan Hydrochloride (including excipients), PPIs, amoxicillin, clarithromycin, metronidazole, levofloxacin, tetracycline, furazolidone, or excipients in 13C-UBT (mannitol, citric acid, or aspartame).
9. History of alcohol abuse, illicit drug use, or drug addiction within 12 months prior to screening, or weekly alcohol intake exceeding 21 units (1 unit = 12 oz/300 ml beer, 1.5 oz/25 ml spirits, or 5 oz/100 ml wine).
10. Use of antibiotics, bismuth agents, or antiprotozoal drugs within 30 days prior to 13C-UBT, or use of H2 receptor antagonists, PPIs, or interfering drugs (e.g., sodium succinate) within 14 days.
11. Concurrent use of drugs contraindicated with clarithromycin (e.g., colchicine, pimozide, ergot derivatives, tadalafil, terfenadine, astemizole, cisapride, simvastatin, lovastatin, atorvastatin, etc.)..Use of pravastatin, fluvastatin, or rosuvastatin is permitted but should be used with caution.
12. Concurrent use of strong CYP2C19 or CYP3A4 inhibitors or inducers (e.g., fluconazole, fluoxetine, fluvoxamine, ticlopidine, rifampin, ritonavir, itraconazole, ketoconazole, indinavir, nelfinavir, saquinavir, telithromycin).
13. History of surgeries affecting gastric acid secretion, such as gastric resection or vagotomy.
14. Significant central nervous, cardiovascular, hepatic, pulmonary, renal, metabolic, gastrointestinal, urological, reproductive, endocrine, or hematological disorders that may affect the study results or participant safety, as judged by the investigator.
15. History of any malignancy, including MALT lymphoma.
16. Need for hospitalization or surgery during the study or within 30 days prior to screening.
17. Diagnosis of AIDS or HIV infection.
18. Female participants who are pregnant, breastfeeding, planning to become pregnant, or planning to donate eggs during the study or within 4 weeks after the study.
19. Participants with negative H. pylori culture during the screening period.
20. Participants with prior P-CAB plus amoxicillin dual therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Successful Eradication of Helicobacter pylori | At least 4 weeks after the last dose of study medication
  The proportion of participants who achieve successful eradication of Helicobacter pylori. Eradication is defined as a negative result on the 13C-Urea Breath Test (13C-UBT) conducted at least 4 weeks after the last dose of the study medication. The eradication rate will be calculated as: Eradication Rate=（Number of Participants with Successful Eradication/ Total number of participants）*100% This outcome will compare the efficacy of Keverprazan Hydrochloride + Amoxicillin dual therapy to susceptibility-guided quadruple therapy in the rescue treatment of H. pylori infection.

IPD SHARING:
Plan to Share IPD: No